CLINICAL TRIAL: NCT03745898
Title: The Impact of Low Flow Nocturnal Oxygen Therapy on Hospital Admissions and Mortality in Patients With Heart Failure and Central Sleep Apnea (LOFT-HF)
Brief Title: The Impact of Low Flow Nocturnal Oxygen Therapy on Hospital Admissions and Mortality in Patients With Heart Failure and Central Sleep Apnea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low feasibility of completion within the study period due to delayed site activation and slow participant accrual
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Susan Redline, Professor and Senior Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U24HL140412-01_UG3; U24HL140412-01 (NIH)
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Central Sleep Apnea
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Central | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nocturnal Oxygen Therapy (Active Comparator): Active nocturnal oxygen therapy
  Interventions: Drug: Oxygen
- Sham Nocturnal Oxygen Therapy (Sham Comparator): Sham nocturnal oxygen therapy (room air)
  Interventions: Other: Room Air

INTERVENTIONS:
Drug: Oxygen — Active nocturnal oxygen concentrator
  Arms: Nocturnal Oxygen Therapy
Other: Room Air — Sham nocturnal oxygen concentrator (room air)
  Other Names: Sham Oxygen
  Arms: Sham Nocturnal Oxygen Therapy

SUMMARY:
The purpose of this trial is to evaluate the long-term effects of Nocturnal Oxygen Therapy (NOXT) on the mortality and morbidity of patients with stable heart failure and a reduced ejection fraction (HFrEF), already receiving optimal guideline-directed medical therapy (GDMT), who have central sleep apnea (CSA).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 21 years at the date of consent.
* History of chronic, stable heart failure with reduced ejection fraction with left ventricular ejection fraction (LVEF) ≤ 50% determined by echocardiography, radionuclide angiography, left ventriculography, or cardiac magnetic resonance imaging, within the year prior to enrollment.
* Central sleep apnea, defined using as an apnea-hypopnea index (AHI) > 15/h with ≥ 50% central events (apnea and hypopneas).
* New York Heart Association (NYHA) Class III or IV, or NYHA Class II with any of the following:

  1. at least one hospitalization for heart failure within the 24 months prior to enrollment or;
  2. a BMI corrected BNP ≥ 300 pg/ml or a corrected NT-proBNP ≥ 1500 pg/ml or;
  3. an ED visit for HF exacerbation where the patient has received an IV diuretic within 12 months of enrollment.
* Treatment with stable, optimized guideline-directed medical therapies (GDMT) according to applicable guidelines in the U.S. and Canada, where stable is defined as the addition of no new class of disease-modifying drug for ≥ 30 days prior to randomization (reasons for intolerance to GDNT must be documented).
* In the investigator's opinion, willing and able to comply with all study requirements.
* Able to fully understand study information and sign an Institutional Review Board (IRB) approved informed consent (including HIPAA authorization in the U.S.).

Exclusion Criteria:

* Current positive airway pressure use or predominantly obstructive rather than central sleep apnea.
* Oxygen saturation < 90% at rest during the day.
* Nocturnal oxygen saturation < 88% for > 5 continuous minutes unaccompanied by apneas or hypopneas.
* Chronic daytime or nighttime use of supplemental oxygen.
* Participants and their bed-partners who currently smoke in the bedroom.
* Severe pulmonary disease requiring continuous home oxygen therapy or the continuous or frequent intermittent use of oral steroids or documented severe chronic obstructive pulmonary disease (COPD) with forced expiratory volume in 1 second (FEV1) < 50%.
* Cardiac surgery, percutaneous coronary intervention, myocardial infarction or unstable angina within the previous 3 months.
* Transient ischemic attack or stroke within the previous 3 months.
* Cardiac resynchronization therapy implantation scheduled or performed within 3 months prior to randomization.
* Primary hemodynamically-significant uncorrected valvular heart disease (obstructive or regurgitant) or any valvular disease expected to require surgery during the trial.
* Acute myocarditis/pericarditis or other cause of potentially reversible cardiomyopathy (e.g., post-partum cardiomyopathy, tachycardia-induced cardiomyopathy), within the previous 6 months.
* End-stage (Stage D) heart failure (HF) requiring continuous outpatient intravenous (IV) inotropic therapy, placement of ventricular assist device, listing for cardiac transplantation, or end-of-life care (e.g. hospice care).
* Pregnancy or of child bearing potential without a negative pregnancy test within 10 days prior to enrollment.
* Life expectancy < 1 year for diseases unrelated to chronic HF.
* Enrolled or planning to enroll in another study that may conflict with protocol requirements or confound subject results in this trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - University of Arizona, Tucson, Arizona
  - Stanford University, Stanford, California
  - Yale School of Medicine, New Haven, Connecticut
  - University of Miami, Coral Gables, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Saint Luke's Mid America Health Institute, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University Hospitals, Highland Hills, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Main Line Health, Wynnewood, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All relevant deidentified data will be deposited in Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) and the National Sleep Research Resource (NSRR)

REFERENCES:
- [Derived] Redline S, Li D, Javaheri S, Patel SR, Parthasarathy S, Fang JC, Brown LK, Dunlap M, Badr MS, Shah N, Chi L, Majid R, Teodorescu M, Stewart G, Hsich E, Polonsky T, Vader J, Johnson MR, Auckley D, Yaggi HK, Kao A, Azarbarzin A, Alex R, Rueschman M, Wolfe L, Gottlieb DJ, Sands SA, Zee PC, Mehra R, Mokhlesi B, Khayat R, Lewis EF, Abraham WT, Wang R. Nocturnal Oxygen Therapy for Central Sleep Apnea in Patients with Heart Failure: A Multisite, Double-Blind, Sham-controlled Randomized Clinical Trial (LOFT-HF). Ann Am Thorac Soc. 2025 Dec;22(12):1951-1960. doi: 10.1513/AnnalsATS.202504-409OC. PMID 40929650

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
Started | 48 | 50
Completed | 48 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Recruitment incomplete due to early termination
Groups:
- Total: Total of all reporting groups
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 28 | 63
  >=65 years | 13 | 22 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.56 (12.22) | 62.78 (11.12) | 61.69 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 36 | 39 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 10 | 28
  White | 29 | 37 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 50 | 98

OUTCOME MEASURES:

1. Primary Outcome: First Occurrence of Mortality Due to Any Cause or an Unplanned Hospitalization for Worsening Heart Failure or a Life-saving Cardiovascular (CV) Intervention
Description: This is a composite primary outcome
Time Frame: 12 months
Population: Recruitment incomplete due to early termination
Measure: Count of Participants; unit: Participants
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
Number analyzed (Participants) | 48 | 50
Participants | 15 | 9

2. Secondary Outcome: Recurrent Event Analyses of Mortality and Morbidity
Description: Count of occurrences of mortality due to any cause or an unplanned hospitalization for worsening heart failure or a Life-saving Cardiovascular (CV) Intervention. (Death, Hospitalization HF / Outpatient HF, Myocardial Infarction / Unstable Angina, Resuscitated Cardiac Arrest, Stroke)
Time Frame: From enrollment to study termination, attrition or death. Min = 41 days, Max = 626 Days
Population: Incomplete due to early termination
Measure: Number; unit: events
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
Number analyzed (Participants) | 48 | 50
events | 22 | 18

3. Secondary Outcome: Quality of Life and Symptoms - HF Disease-specific Quality of Life
Description: HF disease-specific quality of life will be assessed by the change in the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life for those who have heart failure. An overall summary score is derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline, 6 month follow up
Population: Incomplete due to early termination
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
Number analyzed (Participants) | 34 | 38
score on a scale | 7.19 (22.32) | 4.83 (13.43)

4. Secondary Outcome: Quality of Life and Symptoms - Generic-quality of Life
Description: Generic-quality of life will be assessed by the change in the Euroqol - 5 Dimensions (EQ-5D) questionnaire. The questionnaire comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. A total score in calculated using a US-specific weighted algorithm with a possible range [-0.109,1], where 1 represents the best outcome with 'no problems' selected for every item on the scale.
Time Frame: Baseline, 6 month follow up
Population: Incomplete due to early termination
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
Number analyzed (Participants) | 34 | 38
score on a scale | 0.06 (0.19) | 0.02 (0.11)

5. Secondary Outcome: Quality of Life and Symptoms - Depressive Symptoms
Description: Depressive symptoms will be assessed by the change in the Patient Health Questionnaire - 8 items (PHQ-8). A scores ranges from 0 to 24. A score greater than 10 is considered major depression and a score 20 or more is considered severe major depression.
Time Frame: Baseline, 6 month follow up
Population: Incomplete due to early termination
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
Number analyzed (Participants) | 33 | 38
score on a scale | -2.21 (5.01) | -1.61 (5.85)

6. Secondary Outcome: Quality of Life and Symptoms - Sleep Symptoms and Sleep Related Daytime Impairment
Description: Sleep symptoms and sleep related daytime impairment will be assessed by the change in the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (SD) Questionnaire and Sleep Related Impairment (SRI) Questionnaire. The final score for each is represented by the T-score, a standardized score with a population mean of 50 and a standard deviation (SD) of 10, where a higher score indicates a worse score. For SRI a T-score >= 60 implies high levels of sleep related impairment, and for PROMIS SD a T-score >= 60 implies high levels of sleep disturbance.
Time Frame: Baseline, 6 month follow up
Population: Incomplete due to early termination
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
Number analyzed (Participants) | 32 | 37
score on a scale
  Change in Sleep Disturbance Scale T-score | -6.26 (7.77) | -4.98 (8.32)
  Change in Sleep Related Impairment Scale T-score | -5.69 (9.42) | -4.20 (12.62)

7. Secondary Outcome: Functional Status
Description: Functional status will be assessed by the change in New York Heart Association (NYHA) Functional Class Ranking, where higher classes indicate decreased function (worse outcome). Possible Classes are I-IV, which indicate a score of 1-4. Class I indicates No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath. ; Class II indicates Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain. ; Class III indicates Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain. ; and Class IV indicates Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Time Frame: Baseline, 6 month follow up
Population: Incomplete due to early termination
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
Number analyzed (Participants) | 31 | 35
score on a scale | -0.16 (0.52) | -0.03 (0.57)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events from study enrollment through all follow-up study visits (baseline, 3 month, 6 month, 9 month 12 month, 18 month, 24 month) until study termination.
Arm/Group | Nocturnal Oxygen Therapy | Sham Nocturnal Oxygen Therapy
All-Cause Mortality (participants affected / at risk) | 6/48 | 6/50
Serious Adverse Events (participants affected / at risk) | 26/48 | 22/50
Other Adverse Events (participants affected / at risk) | 6/48 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nocturnal Oxygen Therapy (N=48) | Sham Nocturnal Oxygen Therapy (N=50)
2019 novel coronavirus infection (Infections and infestations) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Acute decompensated heart failure (Cardiac disorders) | 4 (5) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angiogram (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Biventricular cardioverter defibrillator replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Bronchitis viral (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 2 (2)
Cardiac catheterization (Investigations) | 2 (2) | 0 (0)
Cardiac death (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker malfunction (Product Issues) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (2) | 0 (0)
Chest pain (General disorders) | 1 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 3 (6) | 4 (4)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cryoablation (Surgical and medical procedures) | 1 (1) | 0 (0)
DC shock (Surgical and medical procedures) | 0 (0) | 1 (1)
Death (General disorders) | 6 (6) | 4 (4)
Decompensated heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic foot ulcer (Endocrine disorders) | 0 (0) | 2 (2)
Diveticulitis intestinal perforated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Vascular disorders) | 0 (0) | 1 (1)
Driver in motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Edema lower limb (Cardiac disorders) | 0 (0) | 1 (1)
Eosinophillic esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Flu (Infections and infestations) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gangrene toe (Infections and infestations) | 0 (0) | 1 (1)
GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2) | 1 (2)
Heart transplant (Surgical and medical procedures) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Implantable cardioverter defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal bleeding (Vascular disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotizing fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Shortness of breath (Cardiac disorders) | 1 (1) | 1 (1)
Sickle cell disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Vascular disorders) | 0 (0) | 2 (3)
Tenotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Volume overload (Cardiac disorders) | 0 (0) | 1 (1)
Weakness (General disorders) | 0 (0) | 1 (1)
Whooping cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nocturnal Oxygen Therapy (N=48) | Sham Nocturnal Oxygen Therapy (N=50)
2019 novel coronavirus infection (Infections and infestations) | 3 (3) | 3 (3)
Congestive heart failure (Cardiac disorders) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Study incomplete due to early termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03745898/Prot_SAP_000.pdf